CLINICAL TRIAL: NCT06378632
Title: An International Multi-center Observational, Single-arm, Blinded Study to Assess the Performance of the Cordio HearO System
Brief Title: AN INTERNATIONAL, OBSERVATIONAL, BLINDED STUDY TO ASSESS THE PERFORMANCE OF THE CORDIO HEARO SYSTEM
Acronym: DETECT-HF
Status: Recruiting | Type: Observational
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0011 DETECT-HF
Record Dates: First submitted 2024-04-14; First posted 2024-04-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Hearo App — No intervention - only data collection

SUMMARY:
Study Design:

This is an international, multicenter, observational, non-interventional, prospective, blinded, single-arm, two-period study, to collect patient utterances that will be retrospectively analyzed to determine the sensitivity and UPNR of the HearO system.

DETAILED DESCRIPTION:
Two periods:

Run-In period will be a period in which patients will submit daily recordings, baseline creation

Core period will be a period in which patients will be followed up and will continually submit daily recordings for up-to 24 months per patient or until End-of-Study (EOS), whichever comes first.

ELIGIBILITY:
Major Inclusion Criteria:

1. Age 22 or greater
2. Diagnosed with Symptomatic Chronic Heart Failure [NYHA II-IVa (ambulatory)]
3. At least one of the following:

   1. One ADHF hospitalization in the last 12 months
   2. One unplanned IV/SC diuretic administration in the last 6 months
   3. Two unplanned IV/SC diuretic administrations in the last 12 months
   4. NTProBNP >500 pg/ml
4. Clinically stable HF according to investigator discretion
5. Willing to participate as evidenced by signing the written informed consent.

Major Exclusion Criteria:

1. Unable to comply with daily use of the App,
2. Has had a major cardiovascular event within 3 months prior to enrolment.
3. Had a Cardiac Resynchronization Therapy Device (CRT) implanted or upgrading ≤ 1 month prior to screening visit.
4. Has estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73.
5. Is likely to undergo heart transplantation/ LVAD within 6 months of Screening Visit.
6. Was treated for a significant COPD

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Events (HFEs) | EOS is defined as when a total of at least 78 first usable and CEC-adjudicated HFEs have occurred or up-to 24 months per patient
  Until the end of the study, each participant will be assigned to one of the following event outcomes:
  1. Having at least one protocol-defined Heart Failure Event (HFE) in the CORE period
  2. Having no Heart Failure Event (HFE) during the entire CORE period

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Haviv, PhD, Study Director — Cordio Medical
Locations (45):
- United States (37):
  - Eastern Shore Research Institute, Fairhope, Alabama
  - UC San Diego Health, La Jolla, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - VA San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Nature Coast Clinical Research, Crystal River, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Amavita Clinical Research, Miami, Florida
  - Advance Medical Research Services Corp (AMRS), Miami, Florida
  - Baptist Health (Miami Cardiac & Vascular Institute), Miami, Florida
  - Comprehensive Medical & Research Center, Plantation, Florida
  - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - Tampa General Hospital, Tampa, Florida
  - West Georgia Cardiology, Carrollton, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Illinois Masonic Health Center, Downers Grove, Illinois
  - Midwest Cardiovascular Center, Naperville, Illinois
  - Robert J. Dole VA Medical Center, Wichita, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Nebraska Heart Center, Lincoln, Nebraska
  - VA Southern Nevada Healthcare System, North Las Vegas, Nevada
  - Mount Sinai Morningside, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Mission Hospital, Asheville, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Rio Grande Regional Hospital, McAllen, Texas
  - Methodist Hospital of San Antonio, San Antonio, Texas
- Israel (7):
  - University Hospital Samson Assuta Ashdod, Ashdod
  - Assuta Be'er Sheva Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galiee Medical Center, Nahariya
  - Tel Aviv Sourasky (Ichilov) Medical Center, Tel Aviv
  - Poriya Medical Center, Tiberias
- Hospital Universitari Germans Trias i Pujol, Badalona, Spain

IPD SHARING:
Plan to Share IPD: No